CLINICAL TRIAL: NCT06603909
Title: Health Outcomes of Nasopharyngeal Carcinoma Patients Three Years After Treatment by the AI-assisted Home Enteral Nutrition Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changsha Medical University (Other)
Responsible Party: Principal Investigator, Danna Chen, Doctor, Changsha Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AI-nutrition to NPC patients
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer, Carcinoma; Artificial Intelligence (AI); Nutrition
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group 1: Use AI to assist nutrition management (Experimental): The first step: Preliminary clinical nutrition screening and evaluation. Information of patients' age, stage of nasopharyngeal cancer, treatment stage (radiotherapy, chemotherapy stage) and other information were collected, and the management plan was determined.
  The second step: AI-assisted HEN management mode. Regular nutritional monitoring and follow-up of patients were conducted by means of intelligent computer, intelligent App body fat device and mobile communication network collection, and basic signs, nutritional status, nutritional risks and implementation of support programs of patients were managed. Nutritional analysis model and index model are used to start the intelligent daily monitoring management and acute attack early warning mechanism.
  The third step: Monitor and alert. The AI system popularized the basic knowledge of nutrition to patients through the App platform.
  Interventions: Other: group 1: Use AI to assist nutrition management
- group 2: Contact the nutritionist team of the hospital for nutrition management (Experimental): Contact the nutritionist team of the hospital for nutrition management according to patients' own situation
  Interventions: Other: group 2：Traditional nutrition management（through the hospital dietitian）
- group 3: Do not adopt the two management methods. (No Intervention): blank control group

INTERVENTIONS:
Other: group 1: Use AI to assist nutrition management — group1：AI-assisted nutrition management. group 2：Traditional nutrition management（through the hospital dietitian）.group 3:control.
  Arms: group 1: Use AI to assist nutrition management
Other: group 2：Traditional nutrition management（through the hospital dietitian） — group 2：Traditional nutrition management（through the hospital dietitian）
  Arms: group 2: Contact the nutritionist team of the hospital for nutrition management

SUMMARY:
You have completed the current stage of cancer treatment, after which you need to check regularly and pay attention to nutrition. So we started this study to see if AI could help with nutrition management. Main options: Option 1: Use AI to assist nutrition management; Option 2: Contact the nutritionist team of the hospital for nutrition management according to your own situation. Option 3: Do not adopt the first two management methods. Special Statement: Please choose; Cancer screening data is used for statistical analysis, but does not reveal any personal privacy.

ELIGIBILITY:
Inclusion Criteria:

* Malignant tumor patient

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Survival Rate | three years after treatment
  Survival Rate
Local Recurrence Rate | three years after treatment
  Local Recurrence Rate

SECONDARY OUTCOMES:
DNA positive rate of Epstein-Barr(EB) virus | three years after treatment
  DNA positive rate of Epstein-Barr(EB) virus
Body mass index | three years after treatment
  Data was obtained through the intelligent body fat device

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Zhengzhou University, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Publish the paper publicly so that more people can learn about the results of the study
Supporting Information: Study Protocol

REFERENCES:
- [Background] Kulkarni S, Seneviratne N, Baig MS, Khan AHA. Artificial Intelligence in Medicine: Where Are We Now? Acad Radiol. 2020 Jan;27(1):62-70. doi: 10.1016/j.acra.2019.10.001. Epub 2019 Oct 19. PMID 31636002
- [Background] Mundi MS, Mohamed Elfadil O, Olson DA, Pattinson AK, Epp LM, Miller LD, Seegmiller SL, Schneckloth JM, Baker MR, Abdelmagid MG, Patel A, Wescott BA, Elder LS, Hagenbrock MC, Sefried LE, Hurt RT. Home enteral nutrition: A descriptive study. JPEN J Parenter Enteral Nutr. 2023 May;47(4):550-562. doi: 10.1002/jpen.2498. Epub 2023 Apr 12. PMID 36912121
- [Background] Bischoff SC, Austin P, Boeykens K, Chourdakis M, Cuerda C, Jonkers-Schuitema C, Lichota M, Nyulasi I, Schneider SM, Stanga Z, Pironi L. ESPEN practical guideline: Home enteral nutrition. Clin Nutr. 2022 Feb;41(2):468-488. doi: 10.1016/j.clnu.2021.10.018. Epub 2021 Nov 24. PMID 35007816
- [Background] Muscaritoli M, Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Oldervoll L, Ravasco P, Solheim TS, Strasser F, de van der Schueren M, Preiser JC, Bischoff SC. ESPEN practical guideline: Clinical Nutrition in cancer. Clin Nutr. 2021 May;40(5):2898-2913. doi: 10.1016/j.clnu.2021.02.005. Epub 2021 Mar 15. PMID 33946039
- [Derived] Liu J, Wang X, Ye X, Chen D. Improved health outcomes of nasopharyngeal carcinoma patients 3 years after treatment by the AI-assisted home enteral nutrition management. Front Nutr. 2025 Jan 7;11:1481073. doi: 10.3389/fnut.2024.1481073. eCollection 2024. PMID 39839291